CLINICAL TRIAL: NCT02433639
Title: Study of TH-302 Monotherapy as Second-line Treatment in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Do-Youn Oh, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1412-023-631
Record Dates: First submitted 2015-04-26; First posted 2015-05-05 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Biliary Tract Cancer
Keywords: advanced biliary tract cancer, TH-302
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): single arm study: TH-302 monotherapy is given
  Interventions: Drug: TH-302 monotherapy

INTERVENTIONS:
Drug: TH-302 monotherapy — TH-302 (480 ) mg/m2 D1, D8, D15 Q 4 weeks

SUMMARY:
Biliary tract cancer is relatively rare cancer, with generally poor prognosis. In metastatic/recurrent biliary tract cancer, the most commonly used 1st-line chemotherapy is gemcitabine+cisplatin combination. However, there is no standard 2nd-line chemotherapy and there is no validated targeted therapeutic agent, even though this tumor harbors diverse genetic characteristics.

TH-302 (1-methyl-2-nitro-1H-imidazole-5-yl)methyl N,N'-bis(2-bromoethyl) diamidophos-phate is a nitroimidazole-linked prodrug of a brominated version of isophosphoramide mustard (Br-IPM). When exposed to hypoxic conditions, TH-302 is reduced at the nitroimadazole site of the prodrug by intracellular reductases leading to the release of Br-IPM. Br-IPM can then act as a DNA crosslinking agent. In areas of normoxia, TH-302 remains intact as a prodrug and toxicity is minimized. In addition, preclinical data suggest that after activation, the active moiety may diffuse to areas outside the hypoxic region, demonstrating a "bystander" effect and possibly exhibiting additional anti-tumor activity.

It is well known that biliary tract cancer is hypovascular tumor, so it contains large hypoxic area in the tumor. Therefore it would be worthy to test TH-302 in biliary tract cancer.

This study is a phase II study of TH-302 monotherapy as second-line treatment in advanced biliary tract cancer, to investigate efficacy and safety of TH-302 monotherapy.

DETAILED DESCRIPTION:
Biliary tract cancer is relatively rare disease worldwide among all kinds of solid tumors. However the incidence of biliary tract cancer is relatively higher in Korea compared to the western countries. The prognosis of all biliary tract cancer is poor, that is, the 5-year overall survival rate is 26.7%. The main reasons of poor prognosis are: 1) there is no screening method to detect in early stage, 2) the relapse rate after curative surgery is high, 3) in metastatic/recurrent biliary tract cancer, the chemo-sensitivity is relatively low. And another important reason of poor prognosis is low interest of investigators. So the researches with new agents have been limited compared with other types of cancer such as lung cancer, breast cancer and colon cancer etc. In metastatic/recurrent biliary tract cancer, the available cytotoxic chemotherapies are composed of gemcitabine, cisplatin, 5-FU, etc. The most commonly used 1st-line chemotherapy is gemcitabine+cisplatin combination. (N Engl J Med 2010; 362 (14): 1273-81) There is no standard 2nd-line chemotherapy so far.

The overall survival with these cytotoxic chemotherapies is about 8-10 months. So far, there is no validated targeted therapeutic agent in biliary tract cancer, even though this tumor harbors diverse genetic characteristics.

Therefore, there is a huge unmet medical need in biliary tract cancer.

TH-302 (1-methyl-2-nitro-1H-imidazole-5-yl)methyl N,N'-bis(2-bromoethyl) diamidophos-phate is a nitroimidazole-linked prodrug of a brominated version of isophosphoramide mustard (Br-IPM). When exposed to hypoxic conditions, TH-302 is reduced at the nitroimadazole site of the prodrug by intracellular reductases leading to the release of Br-IPM. Br-IPM can then act as a DNA crosslinking agent. Tumors often consist of large areas of highly hypoxic regions that are known to be resistant to chemotherapy and radiation treatment. In areas of normoxia, TH-302 remains intact as a prodrug and toxicity is minimized. Thus, TH-302 has been designed to target these highly hypoxic tumor regions and this makes it an attractive candidate for clinical development. In addition, preclinical data suggest that after activation, the active moiety may diffuse to areas outside the hypoxic region, demonstrating a "bystander" effect and possibly exhibiting additional anti-tumor activity.

It is well known that biliary tract cancer is hypovascular tumor, so it contains large hypoxic area in the tumor. Therefore it would be worthy to test TH-302 in biliary tract cancer.

This study is a phase II study of TH-302 monotherapy as second-line treatment in advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically / cytologically verified, non-resectable, recurrent, or metastatic biliary tract carcinoma including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma.
2. Patients who were previously treated with one palliative chemotherapy (patients who recurred within 6 months after completion or during adjuvant chemotherapy are allowed)
3. Patients must have measurable or evaluable disease by RECIST 1.1
4. ECOG PS: 0, 1
5. Age ≥ 20 years
6. Adequate bone marrow function defined as: Hb ≥ 8 g/dl, ANC ≥ 1500/mcL, Platelets ≥ 100K/mcL
7. Adequate renal function defined as serum creatinine < 1.6 mg/dl and/or measured creatinine clearance from 24-hour urine collection of ≥ 60 ml/min
8. Adequate hepatic function defined as total bilirubin ≤ 2 mg/dl, ALT/AST ≤ 5 x ULN.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Evidence of another active cancer that may influence patient outcome, except for nonmelanoma skin carcinoma, melanoma in-situ, in-situ carcinoma of the cervix curatively treated, treated superficial bladder cancer, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable.
2. Known brain metastases or primary central nervous system tumors with seizures that are not well controlled with standard medical therapy.
3. Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements.
4. Known HIV positive patient
5. Significant cardiovascular disease including congestive heart failure (New York Heart Association Class II or higher) or active angina pectoris.
6. History of a myocardial infarction within 6 months.
7. History of a stroke or transient ischemic attack within 6 months.
8. Clinically significant peripheral vascular disease.
9. Major surgical procedure within 4 weeks.
10. Uncontrolled infection.
11. Pregnant (positive pregnancy test)
12. Breast-feeding should be discontinued if a nursing mother is to be treated on clinical trial.
13. History of any organ or bone marrow transplant.
14. Subjects who are taking medications that prolong QT interval and have a risk of Torsades de Pointes.
15. Subjects taking a medication that is a moderate or strong inhibitor or inducer of CYP3A4.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
progression-free survival at 4-months (PFS4mo) | 4 months
  PFS is defined as the interval from the date of enrollment to the date of disease progression or death due to any cause, whichever occurs first. PFS4m is defined as the proportion of patients alive and progression-free at 4 months relative to all enrolled patients.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
Disease Control Rate (DCR) | 6 months
Duration of Response (DR) | 2 years
Progression-Free Survival (PFS) | 2 years
Time to Progression (TTP) | 10 months
Overall Survival (OS) | 2 years
safety and tolerability as measured by number and grade of toxicity events | 15 months
  Overall Safety Profile, as characterized by type, frequency, severity as graded by NCI Common Toxicity Criteria for Adverse Events version 4.0 (NCI CTCAEv4.0), timing and relationship to treatment, and laboratory abnormalities observed.

OTHER OUTCOMES:
protein/genomic biomarkers of efficacy from serum, plasma or tumor | 2 years
  To explore the association of potential predictive biomarkers and of hypoxia biomarkers from serum, plasma, and tumor with efficacy endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea